CLINICAL TRIAL: NCT01295645
Title: A Phase II Randomized Study of Cidofovir Versus Best Supportive Care for Polyomavirus Hominis Type I (BK) Virus Related Hemorrhagic Cystitis After Stem Cell Transplant
Brief Title: Cidofovir Versus Best Supportive Care for Hemorrhagic Cystitis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0518; NCI-2011-00250 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-02-10; First posted 2011-02-14 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Transplantation Infection
Keywords: Stem Cell Transplant; Hemorrhagic Cystitis; Bladder inflammation; Frequent urination; Pain; Polyomavirus hominis type I; BK virus; BKV; Cidofovir; Vistide
MeSH Terms: conditions — Cystitis, Hemorrhagic; Cystitis; Pain | interventions — Cidofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care + Cidofovir (Experimental): Cidofovir 0.5 mg/kg IV 3 x week for 4 weeks
  Interventions: Drug: Cidofovir
- No Cidofovir (Active Comparator): Standard of Care: Pharmacologic management of pain, spasms, and urinary urgency with medications, hyper-hydration, or continuous bladder irrigation.
  Interventions: Other: No Cidofovir

INTERVENTIONS:
Drug: Cidofovir — 0.5 mg/kg by vein (IV) 3 times a week for 4 weeks.
  Other Names: Vistide
  Arms: Standard of Care + Cidofovir
Other: No Cidofovir — Standard of Care: Pharmacologic management of pain, spasms, and urinary urgency with medications, hyper-hydration, or continuous bladder irrigation.
  Arms: No Cidofovir

SUMMARY:
The goal of this clinical research study is to learn if adding cidofovir to the standard of care can improve symptoms of hemorrhagic cystitis caused by the BK virus as compared to standard of care alone. The safety of cidofovir will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

Cidofovir is an anti-viral drug that is designed to treat or prevent infections caused by certain kinds of viruses.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups and you will have an equal chance of being in either group:

* If you are in Group 1, you will receive standard of care drugs and cidofovir. The doctor will tell you more about the standard of care drugs that you will take and the risks for them.
* If you are in Group 2, you will only receive standard of care drugs.

Study Drug Administration:

If you are in Group 1, you will receive cidofovir by vein over about 1 hour 3 times per week. You will also receive standard of care, which may include oral pain drugs taken every 4 to 6 hours as needed, oral drugs for urinary urgency taken 2 times daily, and fluids given by vein to increase your urination rate.

If you are in Group 2, you will only receive the standard of care, as described above.

Study Visits:

Each week:

* Blood (about 2 tablespoons) will be drawn for routine tests.
* You will have a physical exam, including measurement of your vital signs.

Every 2 weeks, you will complete the questionnaire about urinary problems.

Length of Study:

If you are in Group 1, you may continue taking the study drug for up to 4 weeks. Group 2 will take the standard of care for 4 weeks. If the doctor thinks it is needed Groups 1 and 2 can continue to receive standard of care after this study is over. If your symptoms get worse during the study and you are not receiving cidofovir, you may be eligible for further treatments, which may include cidofovir, after the study ends. You will no longer be able to take the study drug if the disease gets worse or intolerable side effects occur.

Your participation on the study will be over once you have completed the end-of-treatment visit and the follow-up visit.

End-of-Treatment Visit:

After you finish treatment:

* Urine will be collected to test the level of BK virus.
* You will complete the questionnaire about urinary problems.

Follow-up Visit:

Four (4) weeks after treatment ends:

* You will have a physical exam, including measurement of your vital signs.
* Urine will be collected to test the level of BK virus.

This is an investigational study. Cidofovir is FDA approved and commercially available for the treatment of several viral infections. Its use in patients with the BK virus after a stem cell transplant is investigational.

Up to 40 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. HSCT patients with symptomatic hemorrhagic cystitis (minimal Grade 1 symptoms of HC per NCI criteria) and positive BKV in urine >1x103 DNA copies/ml
2. Age >/= 6 years
3. Patient must sign the informed consent document.

Exclusion Criteria:

1. Creatine clearance < 55 ml/min, calculated using ideal body weight (IBW) using Cockcroft-Gault equation
2. Concomitant use of foscarnet, liposomal amphotericin B or aminoglycoside
3. Use of cidofovir for bladder instillation
4. Use of formalin or hyperbaric oxygen treatment

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-03-17 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Microbiologic Response | 8 weeks
  Response defined as improvement in symptoms based on questionnaire, reduction or stability in grade of hemorrhagic cystitis, and level of virus must be a 1 log reduction from baseline when the BKV was first diagnosed.

CONTACTS AND LOCATIONS:
Overall Officials: Borje S. Andersson, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org